CLINICAL TRIAL: NCT04499144
Title: A Modified Approach for the Closure of Oral Sinus Communications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Ralph Habib, Principal investigator, University of Siena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODO002
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Surgery Site Fistula
Keywords: Extraction; Oro-antral communication; Oro-antral fistula
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Intervention Model Description: case series of a new surgical design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified buccal flap and subepithelial connective palatal flap (Experimental)
  Interventions: Procedure: modified buccal flap and subepithelial connective palatal flap

INTERVENTIONS:
Procedure: modified buccal flap and subepithelial connective palatal flap — The connective flap was harvested from the deeper area of the palatal mucosa. Pedicle flap dimensions were reported using the periodontal probe. The flap was then rotated to cover the oro antral communication (OAC) area. The rotation could be in mesial or distal direction, related to OAC position and for the convenience of the donor site. The connective palatal flap was sutured to the buccal periostium using mattress sutures.

SUMMARY:
The aim of this study is to describe a modified surgical approach for the closure of oral sinus communications, using a buccal trapezoidal flap combined with a connective pedicle flap rotated from the palate

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of Oro-antral communication
* Patients with adequate radiographic status
* Patients who read and signed the informed consent
* Patients without periodontal disease
* Patients≥18

Exclusion Criteria:

* Pregnancy or breastfeeding patients
* Patients compliance and patients with mental disorders
* Patients with diabetes
* Patients with osteonecrosis
* Patients with head and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Closure of the communication | Day 30
  Clinical observation

SECONDARY OUTCOMES:
Pain and discomfort | Day 30
  These parameters are described using VAS technique

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Habib, Dr., Principal Investigator — University of Siena
Locations (1):
- University of Siena- Department of medical biotechnologies, Siena, Italy